CLINICAL TRIAL: NCT00305539
Title: HECTHOR: A Pilot Multicenter Double-blind Randomised Study of 3 Months Treatment With Humira Added to Steroids in Giant Cell Arteritis
Brief Title: HECTHOR: Humira to Spare Steroids in Giant Cell Arteritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P041203
Record Dates: First submitted 2006-03-21; First posted 2006-03-22 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis; Placebo; Anti-TNF; Multicenter-randomized-trial; Proved GCA according to ACR criteria (HUNDER et al 1990)
MeSH Terms: conditions — Giant Cell Arteritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: adalimumab
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: adalimumab — 40 mg sc / for 3 months
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
Hypothesis: In giant cell arteritis (GCA), a short initial treatment with anti-TNF may allow a faster decrease of steroids dosage and therefore avoid some of the adverse events of steroids.

DETAILED DESCRIPTION:
The protocol consists of a SC injection of adalimumab or placebo every 2 weeks for 10 weeks added to steroids

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* ACR criteria for Giant cell arteritis (HUNDER 1990)
* Positive Temporal artery biopsy
* Plus standard inclusion criteria for Humira protocols

Exclusion Criteria:

* Prednisone treatment for a different disease at a dose >15 mg/day
* Corticoid treatment for GCA more than 10 days
* GCA treatment with prednisone > 1 mg/kg whatever period of time
* GCA treatment with an anti-TNF, MTX, cyclosporine, cyclophosphamide, dapsone or steroid bolus
* Recent, permanent or transient visual loss due to GCA and the presence of any specific visual abnormality (diplopia, hallucination)
* Plus standard exclusion criteria for Humira protocols

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2006-05; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
To determine the influence of an initial treatment of 3 months with adalimumab, 40 mg every other week, in the percentage of patients achieving at 6 months (week 26), a decrease in their corticosteroid treatment to a dose equal or lower than 0,1 mg/kg | 1 year

SECONDARY OUTCOMES:
To determine the influence of an initial treatment of 3 months with adalimumab on the total dose of corticosteroids determined by AUC (area under the curve) | 1 year
To determine the influence of an initial treatment of 3 months with adalimumab on the percentage of patients relapsing at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, MD, PhD, Principal Investigator — Hôpital Bicêtre, APHP, France
Locations (1):
- Hôpital Bicêtre, Le Kremlin-Bicêtre, France

REFERENCES:
- [Derived] Seror R, Baron G, Hachulla E, Debandt M, Larroche C, Puechal X, Maurier F, de Wazieres B, Quemeneur T, Ravaud P, Mariette X. Adalimumab for steroid sparing in patients with giant-cell arteritis: results of a multicentre randomised controlled trial. Ann Rheum Dis. 2014 Dec;73(12):2074-81. doi: 10.1136/annrheumdis-2013-203586. Epub 2013 Jul 29. PMID 23897775